CLINICAL TRIAL: NCT02141048
Title: Evaluation of the Parent Centre's Positive Parenting Skills Training: A Randomised Controlled Trial.
Brief Title: Evaluation of the Parent Centre's Positive Parenting Skills Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: The Parent Centre (Other)
Responsible Party: Principal Investigator, Soraya Lester, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1952 Lester
Record Dates: First submitted 2014-05-12; First posted 2014-05-16 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Parenting Behaviour; Child Behaviour Problems
Keywords: Parenting programme; Randomised controlled trial; South Africa; Positive parenting; Child behaviour problems; Implementation fidelity; Low- and middle-income country

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive Parenting Skills Training (Experimental): Participants assigned to the intervention group will receive the Positive Parenting Skills Training.
  Interventions: Behavioral: Positive Parenting Skills Training
- Wait-list control (No Intervention): Participants assigned to the wait-list control group will receive no intervention for the duration of this trial. Only after the one-year follow-up assessment has been completed will they receive the Positive Parenting Skills Training.

INTERVENTIONS:
Behavioral: Positive Parenting Skills Training — This parenting programme is delivered by facilitators from the Parent Centre. It is intended for any caregivers of children between the ages of 6-12 years. It consists of seven weekly 3-hour sessions, and is group-based. Once the group size reaches 20 or more people sessions are co-facilitated. The first session provides an overview of the programme. The remaining sessions consider topics including: factors that affect child behaviour, understanding children's feelings, building children's self-esteem, assertive parenting, gaining child-co-operation, effective discipline, and problem solving. The programme is knowledge-based and encourages the development of various parenting skills through the inclusion of experiential activities (e.g., role-plays and homework practice).
  Arms: Positive Parenting Skills Training

SUMMARY:
The purpose of this study is to determine whether the Parent Centre's Positive Parenting Skills Training (PPST), a parenting programme being delivered in South Africa, is effective in improving parenting, and child behaviour related outcomes.

DETAILED DESCRIPTION:
The evaluation of the PPST will assess both the fidelity of the intervention's implementation, as well as the outcomes of the programme in a randomised controlled trial. Programme facilitators and intervention group participants will provide data for the former. For the outcome evaluation, two types of participants will be recruited who will provide self-report data: primary caregivers (n = 80) and where possible another adult living in the home with this primary caregiver and their selected child (n = 60). This "other adult" data will serve to verify the primary caregivers' self-report data. Both participants will provide demographic information, and report on parenting behaviour and child behaviour. Their data will be analysed separately in intention to treat analyses and secondary analyses which consider moderators of programme effectiveness.

ELIGIBILITY:
This study will include two types of participants: (1) primary caregivers and (2) another adult. Both have separate eligibility criteria.

Inclusion Criteria:

1. Primary caregivers (the person most responsible for the well-being of a child)

   * Has a child between the ages of 5-12 years
   * Looks after this child for a minimum of four nights a week
   * Indicated interest in the programme and expressed willingness to enrol in the study
2. Another adult in the household (if available)

   * Lives with the index child (selected by the formerly mentioned caregiver) for at least four nights a week

Exclusion Criteria:

(1) Primary Caregiver

- Has already participated in the Parent Centre's Positive Parenting Skills Training or the Parenting and Leadership Training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in levels of poor and positive parenting on the Parenting Scale (PS), from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  The PS is a self-report measure that can be used to assess dysfunctional discipline practices of parents of young children. It has been validated on a sample of parents who had children between the ages of 5-12 years. The scale is comprised of three factors: verbosity, overreactivity and laxness. It consists of 30 items which can be answered on a 7-point scale. Scale anchors vary per question but are essentially parenting mistakes paired with more effective parenting behaviours (e.g., "I often hold a grudge" vs. "things get back to normal quickly").
Change in levels of poor and positive parenting on the Parent Behaviour Inventory (PBI), from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  The PBI is a self-report measure that is suggested to reflect two dimensions of parenting behaviour: (1) hostile/coercive "behaviour which expresses negative affect or indifference toward the child" and could include using physical punishment, threat or coercion to influence child behaviour; and (2) supportive/engaged parenting which reflects parental acceptance of a child through signs of affection, instrumental and emotional support and shared activities. It is suitable for use with parents of children who are young school-age. The PBI consists of 20 items which can be answered on a 5-point Likert-type scale. Scale anchors range from "not at all true" to "very true".
Change in levels of poor and positive parenting on the Parenting Young Children Scale (PARYC) - Setting Limits subscale, from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  The PARYC is a self-report measure which assesses the frequency of engagement with particular parenting behaviours towards children, on a 7-point Likert scale from "not at all" to "most of the time". It also determines whether performing this behaviour is seen as a problem for the parent with response options including either "yes" or "no". This evaluation will only utilise the Settling Limits subscale which consists of 7 items. The convergent validity of the scale is supported.
Change in levels of child problem behaviour on the Eyberg Child Behaviour Inventory (ECBI), from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  The ECBI can be used to assess behaviour problems in children from 2 to 16 years old. It is comprised of 36 items. Each item is assessed on two dimensions; how often it occurs (i.e., frequency) and identification of the behaviour as a problem for the parent. Frequency ratings are answered on a 7-point Likert-type scale ranging from "never occurs" to "always occurs". By summing these answers together one is provided with an overall problem behaviour Intensity Score. Parents when identifying whether a behaviour is a problem for them answer either "yes" or "no" when asked about the particular behaviour. These answers can also be summed to create a total Problem Score. There is ample evidence for the ECBI to be a psychometrically sound measure, demonstrating its validity and reliability in measuring child problem behaviours.
Change in levels of child problem behaviour on the Child Behaviour Checklist (CBCL) - Externalising Problem subscale, from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  Only the Externalising Problem subscale of the CBCL/6-18 school age version will be used in this study. This subscale is made up of 35 items which assess aggressive and rule breaking behaviour. The subscale assesses such behaviours on a three-point Likert-type scale with options ranging from 0 "not true", to 2 "very true". There is strong support for this scale's psychometric properties.

SECONDARY OUTCOMES:
Change in levels of a parent's sense of competence on the Parenting Sense of Competence Scale (PSOC), from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  This measure is a parent self-report. The PSOC's factor structure is composed of two dimensions of parenting self-esteem namely, efficacy and satisfaction. The scale consists of 17 items which can be answered on a 6-point Likert-type scale ranging from "strongly disagree" to "strongly agree." Some of these items are reverse scored. The scale and its respective subscales have demonstrated high levels of internal consistency. The subscale's convergent and divergent validity are also supported.
Change in levels of conflict and closeness in the parent-child relationship on the Child Parent Relationship Scale (CPRS), from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  The CPRS is a self-report which assesses parent's perceptions of the relationships they have with their children (between 3-12 years). It consists of 15 items, which are answered on a 5-point Likert-type scale. The anchors for this scale range from "does not apply" to "definitely applies". The measure has two subscales; a conflict subscale assesses the extent to which a parent feels that their relationship with their child is characterised by negativity, and a closeness subscale which measures the degree to which a parent feels that the relationship with their child is characterised by open communication, warmth and affection. The scale has adequate evidence for reliability and validity, suggesting it is psychometrically sound.
Change in levels of child self-esteem on the Child Health Questionnaire - Self-esteem subscale (CHQ-ES), from baseline to post-assessment, to the one-year follow-up. | Baseline (prior to programme initiation), post-assessment (shortly after programme conclusion), one-year follow-up (one year after programme conclusion).
  The CHQ-ES is a parent-report. The CHQ measures 14 psychosocial and physical concepts, and is designed and normed for use with children between the ages of 5 and 18 years. Only the self-esteem concept will be used in this evaluation. This concept is comprised of 6 items, which parents can answer on a 5-point Likert-type scale ranging from "very satisfied" to "very dissatisfied". The scale determines how satisfied the parent thinks their child is with aspects of themselves and their lives. Internal consistency reliability in two samples (Australian and American) was found to be above α= 0.8 for this subscale.This scale also shows high levels of item discriminant validity.

CONTACTS AND LOCATIONS:
Overall Officials: Soraya N Lester, MPhil, Principal Investigator — University of Cape Town
Locations (1):
- The Department of Psychology and the School of Management Studies, the University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
All baseline, post-test and follow-up data will be shared on request. Please contact the Principal Investigator for access.

REFERENCES:
- [Background] Kane GA, Wood VA, Barlow J. Parenting programmes: a systematic review and synthesis of qualitative research. Child Care Health Dev. 2007 Nov;33(6):784-93. doi: 10.1111/j.1365-2214.2007.00750.x. PMID 17944788
- [Background] Krug EG, Mercy JA, Dahlberg LL, Zwi AB. [World report on violence and health]. Biomedica. 2002 Dec;22 Suppl 2:327-36. Spanish. PMID 12596453
- [Background] Knerr W, Gardner F, Cluver L. Improving positive parenting skills and reducing harsh and abusive parenting in low- and middle-income countries: a systematic review. Prev Sci. 2013 Aug;14(4):352-63. doi: 10.1007/s11121-012-0314-1. PMID 23315023
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- See also: The Parent Centre's website — http://www.theparentcentre.org.za